CLINICAL TRIAL: NCT00567593
Title: Gene Regulation by Thiazolidinediones
Acronym: GReaT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: James Lewis (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, James Lewis, Professor of Medicine and Epidemiology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DK59961; R01DK059961 (NIH)
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Results first posted 2014-05-08 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rosiglitazone (Other): Rosiglitazone; 8mg tablet once a day for 14 days
  Interventions: Drug: Rosiglitazone

INTERVENTIONS:
Drug: Rosiglitazone — 8mg tablet once a day for 14 days
  Other Names: Avandia

SUMMARY:
The purpose of this study is to determine the effect of rosiglitazone on the genes of the colon

DETAILED DESCRIPTION:
The primary aim of the study is to examine the effect of rosiglitazone (Avandia) on gene regulation in colonic epithelium in the absence of pathologic acute and chronic intestinal inflammation. The secondary aims are to determine the effect of rosiglitazone (Avandia) therapy on T cell activation and cytokine expression in the absence of pathologic acute and chronic intestinal inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* Agrees to use a barrier method of birth control for the duration of the study

Exclusion Criteria:

* History of inflammatory bowel disease
* Has taken prescription or over the counter medications in the two weeks prior to enrollment
* History of diabetes, heart failure, angina, hypertension, coronary heart disease, cancer, bleeding disorder, HIV, AIDS
* Fasting LDL >160 mg/dl
* History of smoking in the year prior to enrollment
* Pregnant or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Lewis, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania Clinical and Translational Research Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rosiglitazone
Started | 12
Completed | 10
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Rosaglitazone: Rosiglitazone: 8mg tablet once a day for 14 days
Arm/Group | Rosaglitazone
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: PDK4 mRNA
Time Frame: 14 days
Measure: Median (Full Range); unit: copies/nL
Arm/Group | Rosiglitazone
Number analyzed (Participants) | 10
copies/nL
  Pre-treatment | .776 [.617 to 1.43]
  Post-treatment | 1.30 [.672 to 1.96]
Statistical Analysis 1: Comparison: Rosiglitazone; Test type: Superiority or Other; p = .01, Wilcoxon (Mann-Whitney); Wilcoxon Rank Sum test

ADVERSE EVENTS:
Time Frame: Adverse events were collected at baseline and during follow-up for up to 30 days after the last administration of study drug.
Arm/Group | Rosiglitazone
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rosiglitazone (N=12)
fatigue (General disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (5)
Headache (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tendonitis in R ring finger (Musculoskeletal and connective tissue disorders) | 1 (2)
Slight cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No